CLINICAL TRIAL: NCT00102245
Title: Clinical and Laboratory Investigation of Humans With Informative Iron or Erythroid Phenotypes
Status: Terminated | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 050085; 05-DK-0085
Record Dates: First submitted 2005-01-25; First posted 2005-01-26 (Estimated); Last update posted 2018-02-14 (Actual); Status verified 2017-08-04

CONDITIONS: Hemoglobinopathies; Hemolysis; Iron Deficiency and Overload; Anemias
Keywords: Hemoglobin; Hemoglobinapathies; Human Genome; Recombinant DNA Technology; Sequencing; Erythrocyte
MeSH Terms: conditions — Hemoglobinopathies; Hemolysis; Iron Deficiencies; Anemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
This study will examine blood for factors that may cause or prevent diseases involving iron or red blood cells. Iron is an important nutrient for human health that is needed to produce red blood cells. Red blood cells carry oxygen to body tissues. A better understanding of iron and red blood cells may help lead to better treatment of several diseases including anemia.

Patients of all ages with red cell abnormalities in the following categories may be eligible for this study:

* Diseases with deficiency, overload or maldistribution of iron
* Known red blood cell diseases, such as anemias and hemoglobinopathies
* Red blood cell diseases of unknown cause, such as hemolysis of unknown cause
* Red blood cell abnormalities with no overt clinical disease, such as hereditary persistence of fetal hemoglobin

Participants undergo the following procedures:

* Medical history
* Physical examination
* Standard medical tests related to the individual's iron or red blood cell condition

Blood draw for the following purposes:

* Testing for syphilis and for the hepatitis B and C, HIV, and HTLV-1viruses, and for a pregnancy test for women who can become pregnant
* Research purposes. This blood is analyzed for genes, proteins, sugars, and fat molecules.

DETAILED DESCRIPTION:
Studies of iron and erythroid cells, have provided fundamental insights into structure function relationships of proteins, energy metabolism, and the molecular basis of many diseases. Based upon the importance of iron for hemoglobin production, the regulation of erythropoiesis and iron metabolism are closely linked, and iron deficiency anemia remains as one of the most common diseases worldwide. The discovery of sickle hemoglobin as having an abnormal electrophoretic mobility marked the beginning of the molecular medicine era. The advent of recombinant DNA technology and sequencing methodologies resulted in the characterization of erythroid cells well beyond that of protein based studies to include gene structure and expression. Globin gene research, in particular, has provided a wealth of information about the expression, regulation and insulation of mammalian genes. More recently, studies of iron absorption and trafficking provided new avenues of research aimed toward growth and energy homeostasis. Genome based approaches were also utilized for the discovery of direct relationships between erythroid cell biology and iron homeostasis. Hence, there is strong evidence that fundamental clinical advances in the field of iron and erythroid biology have been based upon the careful study of humans with informative phenotypes. Clinically based correlation of genotype and phenotype is a proven, systematic approach for understanding the molecular basis of disease.

With the completion of the sequencing of the human genome, a more complete, genetically based description of disease is now achievable. Efforts aimed toward haplotype mapping will further enhance genotype phenotype correlation directly from clinical samples. Considerable progress has already been made in this regard using normal human erythroid cells. In contrast to classic studies involving single genes or proteins, computational biology and high throughput technologies permit the analysis of complex erythroid phenotypes including those with related iron pathologies. This information will be invaluable for understanding those molecular mechanisms that are altered in disease states.

The immediate aim of this protocol is to perform phenotypic analyses in humans with informative iron or erythroid phenotypes. These studies are expected to result in detailed clinical phenotyping and the collection and banking of clinical specimens for further study. In addition, we predict an ongoing growth of new technologies that may eventually be used for molecular and genetic phenotyping of clinical samples (examples include oligonucleotide chips and high throughput mass spectroscopy). Based upon this prediction, we plan to use the samples collected here to assess possible clinical uses of those technologies as they become available. The eventual aim is the discovery of identifiers that may be predictive of disease pathogenesis, severity or clinical response to intervention.

ELIGIBILITY:
* INCLUSION CRITERIA:

A clinically definable iron or erythroid cell phenotype as defined by:

Group 1: Patients with known iron or erythroid diseases (examples: iron deficient anemia or ineffective erythropoiesis).

OR

Group 2: Patients with diseases of unknown etiology (example: unexplained iron overload or anemia).

OR

Group 3: Patients with an informative phenotype in the absence of overt clinical disease (example: hereditary persistence of fetal hemoglobin).

OR

Group 4: Healthy volunteers whose blood or bone marrow samples will be utilized to understand normal iron and erythroid biology and for comparison with the other groups described above.

AGE AND GENDER CONSIDERATIONS:

* Age range: Infancy to unlimited
* Adults: Adults who fall into Groups 1-4 are eligible to enroll in this protocol. They must possess the ability to comprehend the investigational nature of the study and provide informed consent.
* Minors: Minors who fall into groups 1-4 are eligible to enroll in the study for collection of research blood. Within Group 4 (healthy volunteers, minors), the research will not involve greater than minimal risk.

GENERAL EXCLUSION CRITERIA:

Healthy volunteers and Subjects with iron or erythroid diseases who are unable to comprehend the investigational nature of the laboratory research are ineligible to enroll in this protocol.

INCLUSION AND EXCLUSION CRITERIA FOR BONE MARROW SAMPLING:

With the exception of minors, pregnant females, and breast-feeding mothers, volunteers who meet the General Inclusion Criteria for blood collection may be offered the option of bone marrow sampling as part of this protocol. Minors, pregnant females, and breastfeeding mothers will be excluded from bone marrow sampling specifically performed for this protocol. However, they will be asked to consent for collection of up to an additional sample of bone marrow if 1) they are undergoing a bone marrow sampling procedure for clinical purposes, and 2) collection of the additional bone marrow undergoing a clinical procedure if the research sample collection doesn t alter the clinical procedure.

Other bone marrow sampling exclusion criteria include: 1) allergy to xylocaine (lidocaine) or the skin cleansing medication chlorhexidine/Hibiclens. 2) clotting disorders, low platelets (<50,000k) or are taking medications that interfere with blood clotting, such as aspirin, non-steroidal anti-inflammatory agents (such as Motrin or Advil) or blood thinning agents (such as coumadin/warfarin).

Min Age: 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 334 (Actual)
Dates: Start 2005-01-18; Study Completion 2017-08-04

CONTACTS AND LOCATIONS:
Overall Officials: Jeffery L Miller, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Goh SH, Josleyn M, Lee YT, Danner RL, Gherman RB, Cam MC, Miller JL. The human reticulocyte transcriptome. Physiol Genomics. 2007 Jul 18;30(2):172-8. doi: 10.1152/physiolgenomics.00247.2006. Epub 2007 Apr 3. PMID 17405831
- [Background] Gubin AN, Njoroge JM, Wojda U, Pack SD, Rios M, Reid ME, Miller JL. Identification of the dombrock blood group glycoprotein as a polymorphic member of the ADP-ribosyltransferase gene family. Blood. 2000 Oct 1;96(7):2621-7. PMID 11001920
- [Background] Gubin AN, Njoroge JM, Bouffard GG, Miller JL. Gene expression in proliferating human erythroid cells. Genomics. 1999 Jul 15;59(2):168-77. doi: 10.1006/geno.1999.5855. PMID 10409428
- [Background] Miller JL. Signaled expression of fetal hemoglobin during development. Transfusion. 2005 Jul;45(7):1229-32. doi: 10.1111/j.1537-2995.2005.00182.x. No abstract available. PMID 15987371
- [Background] Goh SH, Lee YT, Bhanu NV, Cam MC, Desper R, Martin BM, Moharram R, Gherman RB, Miller JL. A newly discovered human alpha-globin gene. Blood. 2005 Aug 15;106(4):1466-72. doi: 10.1182/blood-2005-03-0948. Epub 2005 Apr 26. PMID 15855277